CLINICAL TRIAL: NCT01300520
Title: The Development of a Surgical Localizing Aid Medical Device and the Determination and Analysis of Significant Variables
Brief Title: The Development of a Surgical Localizing Aid Medical Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough surgeon use to validate the usefulness of the device
Sponsor: Aeos Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TT-1
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Femoral Fracture; Tibial Fracture
Keywords: Fluoroscopy; Femoral fracture; Tibial fracture; Spinal Fusion
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Target Tape (No Intervention): Including target tape in the procedure
- Control (Other): Without target tape in the procedure
  Interventions: Device: Target Tape

INTERVENTIONS:
Device: Target Tape — Comparing procedures using Target Tape against procedures not using Target Tape
  Arms: Control

SUMMARY:
The current method of incision localization in many surgical procedures requires a doctor to reference a medical image, such as an X-ray, to judge where on the body an incision should be made. However, the precise information of the scan is not shown on the patient's skin. Surgeons commonly use palpation to locate the point of incision. They may feel for the area directly or find landmarks under the skin and estimate the location from there. The following factors further complicate palpation: overweight patients, foreign bodies that are difficult to feel for under the skin, fractures with little displacement, or locations under dense muscles. These difficulties are compounded for new surgeons, since palpation is a skill derived through experience.

In many circumstances the surgeon only needs to know where to insert the tool or place the incision - they do not necessarily need to know the depth of the area of interest. If palpation proves ineffective, they may be forced to use fluoroscopy. By referencing the fluoroscopy image the surgeon moves a radiopaque marker, such as their surgical tool, closer to the area of interest. Fluoroscopy is time-consuming, and exposes medical personnel and the patient to radiation. Many fluoroscopic images may be required in a single procedure.

By identifying the efficacy of this new medical device, "Target Tape", there is the potential outcome of making smaller incisions, faster localization, a reduction in fluoroscopy use and a reduced chance in surgical error and the associated costs.

Target Tape is a non invasive device that is in a grid or ruler format that is placed against the subject's skin. The grid/ruler pattern will then appear on the medical imaging scan. Standard surgical skin ink is then used to place these markings in a defined pattern on the skin. This pattern mimics the Target Tape grid or ruler pattern. The medical practitioner can correlate these skin markings to the medical scan image to make their incisions in more accurate locations.

DETAILED DESCRIPTION:
Consent must first be obtained from the prospective patient before Target Tape can be incorporated into the procedure. When a target procedure is scheduled to occur, the surgeon will first determine if Target Tape would be appropriate to use. The procedure will need to be able to integrate Target Tape into it using the Method of Use described above. The decision to then pursue the procedure will be under the discretion of the medical practitioner and consent from the patient. Depending on the procedure, the medical practitioner may need to communicate to the OR or the radiology department to integrate Target Tape into their protocol, since the practitioner making the incisions(s) may not always be the one applying it. Examples of procedures that may utilize Target Tape may be stabilization of fractures, interlocking screw insertions during tibia or femur nailings, breast biopsies, foreign body removals, thoracic and spinal surgeries. Once the procedure is determined to be appropriate to accommodate Target Tape, the medical practitioner will approach the prospective patient and explain how the device will be utilized, the benefits and potential risks associated with it, and answer any questions the patient may have. A representative from Aeos Biomedical may be on hand to aid with this process and may also observe said procedure to record the necessary information. The consent form will then be signed and Target Tape will then be utilized during the procedure.

The methodology of creating an outcome measure will occur over 2 stages with multiple steps in each stage:

Stage I: Proof of Concept

1. Specify measurement goals
2. Proof of Concept Testing
3. Item generation
4. Item reduction

Stage 2: Verification 5. Verification Testing 6. Reliability 7. Validity 8. Interpretability

(i) Subjects (ii) Involved Groups (iii) Data Collection (iv) Statistics

6) Statistical Analysis Sample size

Stage 1:

3 Orthopaedic surgeons, up to 10 patients, per procedure type

3 Spinal surgeons up to 10 patients, per procedure type

3 Plastic surgeons up to 10 patients, per procedure type

2 Thoracic surgeons up to 5 patients, per procedure type

2 Radiologists up to 10 patients, per procedure type

The number of medical practitioners in each type of procedure may fluctuate. Furthermore, this is not a definitive list of specialties. It is foreseeable that a greater variety of procedures from other specialties may be included in the proof of concept testing. Moreover, the number of patients may vary depending on the relative magnitude of the observations and feedback from the medical practitioners.

Stage 2:

The sample sizes for each segment of this stage corresponds to sample sizes used to create outcome measures in the different populations. After Stage 1 has been completed, the sample sizes for Stage 2 will be assessed and a statistical model will be created at that time. A preliminary estimate would require 5 times the sample size per procedure within Stage 1 to be a sufficient.

Variable generation - There is no statistical analysis at this step. It is anticipated that up to 10 procedures would have used the device with at least two different doctors.

Variable reduction - The list of items generated in the step above will be administered to doctors who will be asked to rate the items according to importance. Any items that are deemed insignificant will be removed from the list.

Verification Testing It is anticipated that 5 times the sample size for each procedure will occur in this step. Subject to the testing results of Stage 1, there will be a set of significant performance variables determined for each respective target procedure. Target Tape would then be randomly utilized in the procedures, with controls for who is performing the procedure and patient characteristics. Observation of the significant performance variable occurs for all the procedures

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing a radiological imaging, such as planar X-ray, fluoroscopy, CT or MRI

Exclusion Criteria:

* Subjects who may have allergies to medical skin adhesives, medical skin inks or copper metal

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incision Length | one year
  Measuring the reduction in incision length from using Target Tape

SECONDARY OUTCOMES:
Reduction in Fluoroscopy Exposure | one year
  Measuring the decreased amount of fluoroscopy radiation exposed to the medical staff and the patient.
Procedure Time Savings | One Year
  Measuring the time savings of using Target Tape during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Blachut, MD, FRCS(C), Principal Investigator — The University of British Columbia Department of Orthopaedics
Locations (1):
- The University of British Columbia Department of Orthopaedics, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Margarido CB, Mikhael R, Arzola C, Balki M, Carvalho JC. The intercristal line determined by palpation is not a reliable anatomical landmark for neuraxial anesthesia. Can J Anaesth. 2011 Mar;58(3):262-6. doi: 10.1007/s12630-010-9432-z. Epub 2010 Dec 3. PMID 21128128
- [Background] Benzel, Edward. Spine Surgery: Techniques, Complication, Avoidance, and Management. 2nd. Philadelphia: Elsevier, 2005. 1521-1528. Print
- [Background] Gugala, Zbigniew, Arvind Nana, and Ronald Lindsey.
- [Background] Soar J, Peyton J, Leonard M, Pullyblank AM. Surgical safety checklists. BMJ. 2009 Jan 21;338:b220. doi: 10.1136/bmj.b220. No abstract available. PMID 19158173